CLINICAL TRIAL: NCT05492253
Title: Effect of First Complementary Foods on the Infant Gastrointestinal Microbiota: A Pilot Study
Brief Title: First Complementary Foods and the Infant Gastrointestinal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: American Society for Nutrition Foundation (Unknown)
Responsible Party: Principal Investigator, Jill Trabulsi, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1889964-1
Record Dates: First submitted 2022-07-26; First posted 2022-08-08 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants; Infants; Gastrointestinal Microbiota
Keywords: Healthy term infant; Complementary diet; Gastrointestinal microbiota

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infant cereal (Active Comparator): Oatmeal cereal
  Interventions: Other: Infant grain
- Infant fruit (Experimental): Pureed prunes
  Interventions: Other: Infant fruit
- Infant vegetable (Experimental): Pureed carrots
  Interventions: Other: Infant vegetable
- Infant meat (Experimental): Pureed beef
  Interventions: Other: Infant meat

INTERVENTIONS:
Other: Infant fruit — Infants will be fed prune puree
  Arms: Infant fruit
Other: Infant vegetable — Infants will be fed carrot puree
  Arms: Infant vegetable
Other: Infant meat — Infants will be fed beef puree
  Arms: Infant meat
Other: Infant grain — Infants will be fed oatmeal cereal
  Arms: Infant cereal

SUMMARY:
This study evaluates the effect of different complementary foods on the gastrointestinal microbiota of exclusively human milk fed infants.

DETAILED DESCRIPTION:
The introduction of solid foods plays a role in shaping the microbial communities of the gastrointestinal microbiota. This randomized, controlled, single-blinded trial will evaluate the effect of four infant foods (oatmeal cereal, carrot puree, prune puree, beef and gravy puree) on the gastrointestinal microbiota of exclusively human milk fed infants that have not previously consumed solid foods and who are developmentally ready for the introduction of solid foods.

ELIGIBILITY:
Inclusion Criteria:

* Infant was born vaginally
* Infant was born full term
* Infant has no significant gastrointestinal medical issues/diagnoses (e.g., gastroesophageal reflux, malabsorption syndromes, Celiac disease, Crohn's disease, or physician diagnosed or suspected food allergies)
* Infant is at least 5 months old, but not 8 or more months old
* Infant consumes an exclusively human milk liquid diet only
* Infant has not yet begun consuming solid foods
* Infant is developmentally ready to begin consuming solid foods (i.e., has good head and neck control, can sit upright when supported, and has at least doubled their birth weight)
* Infant has not had antibiotics within the past month
* Infant's nursing mother has not had antibiotics within the past month
* Parent/legal guardian is at least 18 years old

Exclusion Criteria:

* Infant is not developmentally ready to begin solid foods
* Infant has a family history of food allergy

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal microbiota | Day 0, 3, 7, 10, 14
  Composition of the gastrointestinal microbiota (family, genus, and species levels via shotgun metagenomic sequencing) before and after the introduction of solid food

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Trabulsi, PhD, RD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No